CLINICAL TRIAL: NCT07369115
Title: Intra-Cellular Therapies, Inc. / "A Randomized, Double-blind, Placebo-controlled, Single Site Study to Evaluate the Efficacy of Lumateperone for the Treatment of Major Depressive Disorder (MDD) and Early Life Trauma in Adult Patients Aged 21 to 70 Years
Brief Title: Neurocircuitry Mechanisms and Efficacy of Lumateperone as Adjunctive Therapy for Major Depressive Disorder and History of Early Life Abuse
Acronym: ITI-ELA-MDD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Julie Farrington, Clinical Trials Director, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study00008399
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Diorder; Early Life Trauma
MeSH Terms: interventions — lumateperone

STUDY DESIGN:
Intervention Model Description: One group will receive the drug Lumateperone, and the other will receive a placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Drug Arm - Lumateperone (Active Comparator): Lumateperone, 42 mg, for 6 weeks to be taken orally once daily for 25 participants
  Interventions: Drug: Lumateperone 42 mg
- Inactive Drug Arm - Placebo (Placebo Comparator): 25 Participants will receive a matching placebo capsule for 6 weeks to be taken orally once daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lumateperone 42 mg — Lumateperone, 42 mg, will be orally taken by participants once daily for 6 weeks.
  Arms: Active Drug Arm - Lumateperone
Other: Placebo — A matching placebo will be taken orally by participants once daily for 6 weeks.
  Arms: Inactive Drug Arm - Placebo

SUMMARY:
The purpose of this clinical research study is to understand how effective and safe an investigational study drug called lumateperone is and whether it works to reduce the severity of depressive symptoms in adults with Major Depressive Disorder (MDD) and early life trauma. The main questions it aims to answer are:

Aim 1: To assess the efficacy of lumateperone 42 mg administered once daily compared with placebo in the treatment of patients with Major Depressive Disorder and early life abuse.

Aim 2: To assess neurocircuitry encoding of threat and reward learning as predictors of lumateperone response and as mechanisms of treatment action, and assess the change from pre-dose to post-dose of task-evoked brain activation.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before the initiation of any study-specific procedures.

   NOTE: Patients who are unable to independently provide informed consent will be ineligible to participate in this study.
2. Male or female, between the ages of 21 and 70 years, inclusive;
3. Meets the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, Text Revision (DSM-5-TR) criteria for Major Depressive Disorder (MDD) without psychotic symptoms, as confirmed by a trained rater using the modified Structured Clinical Interview (DIAMOND) for DSM-5,
4. MADRS total score ≥ 22 at Screening (Visit 1) and Baseline (Visit 2)
5. Endorse >=1 physical or sexual assault prior to age 16 on the interview-based trauma assessment.

   Many studies refer to early life trauma as prior to age 18. Here we define early life assault as less than 16, rather than 18, in order to ensure a clearer separation between early life and adulthood. While another option might be to restrict even further (e.g., age of trauma < 10), for feasibility (e.g., facilitating recruitment) and generalizability (e.g., results extend to MDD and early life trauma more broadly than just early childhood trauma), we decided on physical or sexual assault prior to age 16.

   Regarding the focus on physical or sexual assault, there are two main reasons. First, the definition of physical and sexual assault can more easily be operationalized through a behavioral description of an event (e.g., has anyone hit you with a fist, has anyone hit you with an object, etc), enabling more precise assessment and detection. Second, there is a robustly elevated risk for mood disorders following assaultive traumas relative to non-assaultive traumas. As such, there is greater clinical need to establish adjunctive treatments among those experiencing assaultive traumas.
6. Participants must have been treated with the same dose of antidepressant therapy for at least 6 weeks, with less than 50% improvement, and be committed to stay on the same stable dosing regimen for the Screening period and for the entire study, at or above the minimally adequate dose in the ATRQ. Documentation of stable and ongoing ADT must be verified by documentation from the subject's psychiatrist, pharmacist, primary care physician, or other qualified healthcare professional.
7. Females of childbearing potential agree to use at least an acceptable method of birth control (including but not limited to hormonal contraception, intrauterine device, vasectomized partner, bilateral tubal occlusion, condom with or without spermicide, cap with spermicide, diaphragm with spermicide, sponge with spermicide, or double barrier methods) from the time informed consent is provided through the end of the SFU period. NOTE: Females of non-childbearing potential (defined as either permanently sterilized, or post-menopausal females [defined as at least one year with no menses without an alternative medical explanation]) are exempt from the birth control requirement.
8. Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

1. Has a current primary DSM-5-TR psychiatric diagnosis other than Major depressive disorder. These include: PTSD, OCD, Bipolar Disorder, Schizophrenia, schizoaffective disorder, or other psychotic disorder. Intellectual disability, Dementia or other cognitive disorders. Moderate or severe substance use disorder (excluding for nicotine)
2. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during the course of his/her participation in the study or

2a. At Screening (Visit 1), the patient scores "yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS within 6 months prior to Screening; or

2b. At Screening (Visit 1), the patient has history of suicidal attempt(s) within 1 year prior to Screening (Visit 1); or

2c. At Baseline/randomization (Visit 2), the patient scores "yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS since the Screening Visit; or

2d. At Screening (Visit 1) or Baseline (Visit 2), scores ≥ 4 on Item 10 (suicidal thoughts) on the rater administered MADRS; or

2e.Considered to be an imminent danger to himself/herself or others.

3. MRI contraindications: History of shrapnel or other metal or electronic implants in the body(such as pacemakers, aneurysm clips, ferrous surgical devices, metallic tattoos on the head, etc.). The patient has received electroconvulsive therapy (ECT), vagal nerve stimulation, or repetitive trans-cranial magnetic stimulation within the past 1 year;

4. The patient has known hypersensitivity or intolerance to lumateperone, or to any of the excipients

5. Treatment with a depot/long-acting injectable antipsychotic within 1 cycle before Screening (Visit 1)

6. The following agents are excluded and must be discontinued at Screening (Visit 1):

6a. Any moderate or strong cytochrome P450 3A4 inhibitor (CYP3A4), or any CYP3A4 inducer 6b. Central opioid agonists/antagonists, including tramadol 6c. Central opioid agonists/antagonists, including tramadol 6d. Dietary supplements and medical foods unless approved by the Sponsor or designee. Daily multivitamin use is permitted

7. Monoamine oxidase inhibitors within 14 days prior to Baseline/Randomization (Visit 2)

8.Other drugs with known psychotropic properties or any non-psychotropic drugs with known or potentially significant central nervous system.

9. The patient plans to initiate psychotherapy or make changes to existing psychotherapy during the study (patients who are participating in stable psychotherapy or psychotherapy as a part of their treatment are allowed to enroll);

10. The patient has participated in a previous clinical trial with lumateperone, or has had exposure to any investigational product within 6 months of the baseline visit or participated in > 2 clinical studies of an investigational product with a central nervous system indication.

11. The patient is pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum pregnancy test at Screening (Visit 1). On Day 1 (Baseline/Visit 2), female patients of childbearing potential must have a negative urine pregnancy test prior to study drug administration;

12. The patient has a positive test for alcohol or drugs of abuse (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, or opioids/opiates) at Screening (Visit 1).

13. The patient has abnormal laboratory values or clinical findings at Screening (Visit 1) including, but not limited to:

13a. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 × the upper limit of normal (ULN) 13b. Total bilirubin > 1.0 × ULN 13c. Hemoglobin < 8 g/dL (80 g/L) for females and < 9 g/dL (90 g/L) for males 13d. Absolute neutrophil count (ANC) < 1200 cells/μL (1.2 × 109 cells/L); 13e. Thyroid-stimulating hormone (TSH) outside of normal reference range AND free T3 or free T4 outside of the reference range. Free T3 and Free T4 will only be evaluated if TSH is outside of reference range; 13f. Poorly controlled diabetes as defined by a glycosylated hemoglobin (HbA1c) >7.5%, despite standard care [> 58 mmol/mol]; 13g. Positive test for hepatitis B surface antigen and/or hepatitis B core antibody immunoglobulin M at screening; positive hepatitis C antibody at Screening (Visit 1), with the exception of a patient for whom the reflex HCV RNA test is negative; 13h. Any other clinically significant abnormal laboratory result obtained at screening (Visit 1)

14. ECG abnormalities where the patient has corrected QT interval using the Fridericia formula (QTcF) > 450 msec for males or > 470 msec for females and/or heart rate < 50 bpm, or evidence of clinically significant bundle-branch blocks at Screening (Visit 1)

15. The patient has any of the following conditions:

Cardiac: uncontrolled angina, or history of a myocardial infarction within 3 months prior to screening, or history of a clinically significant cardiac arrhythmia including antipsychotic drug-induced corrected QT interval prolongation, or any other cardiac disorder;

Malignancy: Any diagnosis of cancer (except basal or squamous cell skin carcinoma), unless in remission for at least 5 years;

Gastrointestinal: history of gastric bypass or any other condition that results in malabsorption;

Endocrine: hypo- or hyperthyroidism unless treated and stable with no medication changes for at least three months prior to screening, diabetes, unless considered stable with no changes in treatment for at least three months prior to screening;

Hepatic: Hepatitis B or Hepatitis C; moderate or severe hepatic impairment (Child-Pugh B or C);

Pulmonary: history of diagnosed and untreated obstructive sleep apnea;

Neurological: history of epilepsy, seizure or convulsion, or electroencephalogram with clinically significant abnormalities, delirium, dementia, amnestic, or central sleep apnea, or significant brain trauma, or other cognitive disorder; History of movement disorders.

Infectious: History of human immunodeficiency virus (HIV) infection.

Note: Any other medical condition, or medical conditions that are stable with treatment (eg, hypertension, hypercholesterolemia, or thyroid abnormalities) are allowed as long as the condition has been stable for at least 3 months prior to Screening (Visit 1); treatments for these conditions are documented, kept stable, and are expected to be unchanged during the study; and the condition is not thought to affect safe participation in the study or relevant study outcomes in the opinion of the Investigator.

16. The patient is judged by the Investigator to be inappropriate for the study;

17. Patient is homeless;

18. Patient does not speak english;

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the absolute change in Montgomery-Åsberg Depression Rating Scale (MADRS) total scores from Baseline to end of Treatment visit at Week 6 in subjects on ADT plus Lumateperone or matching placebo. | Change from Baseline MADRS score at enrollment to end of study (week 7)
  The MADRS is a 10-item questionnaire with each item scored between 0 and 6, resulting in a total score between 0 and 60, with scores above 34 indicating severe depression. Higher MADRS scores indicate more severe depression. The questionnaire is most frequently used in clinical studies to measure outcomes in antidepressant efficacy studies. This scale exhibits construct validity (internal homogeneity) and the concepts of endogenous and non-endogenous depression. The questionnaire includes questions on the following symptoms: (1) apparent sadness; (2) reported sadness; (3) inner tension; (4) reduced sleep; (5) reduced appetite; (6) concentration difficulties; (7) lassitude; (8) inability to feel; (9) pessimistic thoughts; (10) suicidal thoughts. The MADRS must be administered using the Structured Interview Guide for the MADRS (SIGMA). The MADRS total score at screening is a major inclusion criterion of the study, as well as the primary outcome measure for the study.

SECONDARY OUTCOMES:
The key secondary efficacy endpoint is the change from baseline to end of Week 7 in the Clinical Global Impression of Severity (CGI-S) score. | From enrollment to end of study at 7 weeks
  The CGI-S measures the severity of the disease using a 7-point Likert scale ranging from 1=normal, not at all ill to 7=among the most extremely ill subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Health Discovery Building, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernick DM. Stapedectomy results in a residency training program. Ann Otol Rhinol Laryngol. 1986 Sep-Oct;95(5 Pt 1):477-9. doi: 10.1177/000348948609500508. PMID 3767219
- [Background] van Buuren, S., & Groothuis-Oudshoorn, K. (2011). mice: Multivariate Imputation by Chained Equations in R. Journal of Statistical Software, 45(3), 1-67. https://doi.org/10.18637/jss.v045.i03
- [Background] Waddell L, Taylor M. A new self-rating scale for detecting atypical or second-generation antipsychotic side effects. J Psychopharmacol. 2008 May;22(3):238-43. doi: 10.1177/0269881107087976. PMID 18541624
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Guy W (ed). ECDEU Assessment Manual for Psychopharmacology. Clinical Global Impressions (CGI). 1976. Rockville, MD: U.S. Department of Health and Human Services, Public Health Service, Alcohol Drug Abuse and Mental Health Administration, NIMH Psychopharmacology Research Branch, pp. 218-222.
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] First MB, Williams JBW, Benjamin LS, Spitzer RL: User's Guide for the SCID-5-PD (Structured Clinical Interview for DSM-5 Personality Disorder). Arlington, VA, American Psychiatric Association, 2015
- [Background] Chandler GM, Iosifescu DV, Pollack MH, Targum SD, Fava M. RESEARCH: Validation of the Massachusetts General Hospital Antidepressant Treatment History Questionnaire (ATRQ). CNS Neurosci Ther. 2010 Oct;16(5):322-5. doi: 10.1111/j.1755-5949.2009.00102.x. PMID 19769599
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Meltzer HY, Huang M. In vivo actions of atypical antipsychotic drug on serotonergic and dopaminergic systems. Prog Brain Res. 2008;172:177-97. doi: 10.1016/S0079-6123(08)00909-6. PMID 18772033
- [Background] Meltzer HY. The role of serotonin in antipsychotic drug action. Neuropsychopharmacology. 1999 Aug;21(2 Suppl):106S-115S. doi: 10.1016/S0893-133X(99)00046-9. PMID 10432496
- [Background] Hiser J, Heilicher M, Botsford C, Crombie KM, Bellani J, Azar A, Fonzo G, Nacewicz BM, Cisler JM. Decision-making for concurrent reward and threat is differentially modulated by trauma exposure and PTSD symptom severity. Behav Res Ther. 2023 Aug;167:104361. doi: 10.1016/j.brat.2023.104361. Epub 2023 Jun 28. PMID 37393833
- [Background] Weaver SS, Kroska EB, Ross MC, Sartin-Tarm A, Sellnow KA, Schaumberg K, Kiehl KA, Koenigs M, Cisler JM. Sacrificing reward to avoid threat: Characterizing PTSD in the context of a trauma-related approach-avoidance conflict task. J Abnorm Psychol. 2020 Jul;129(5):457-468. doi: 10.1037/abn0000528. Epub 2020 May 21. PMID 32437204
- [Background] Moughrabi N, Botsford C, Gruichich TS, Azar A, Heilicher M, Hiser J, Crombie KM, Dunsmoor JE, Stowe Z, Cisler JM. Large-scale neural network computations and multivariate representations during approach-avoidance conflict decision-making. Neuroimage. 2022 Dec 1;264:119709. doi: 10.1016/j.neuroimage.2022.119709. Epub 2022 Oct 22. PMID 36283543
- [Background] Ironside M, Amemori KI, McGrath CL, Pedersen ML, Kang MS, Amemori S, Frank MJ, Graybiel AM, Pizzagalli DA. Approach-Avoidance Conflict in Major Depressive Disorder: Congruent Neural Findings in Humans and Nonhuman Primates. Biol Psychiatry. 2020 Mar 1;87(5):399-408. doi: 10.1016/j.biopsych.2019.08.022. Epub 2019 Sep 6. PMID 31672243
- [Background] Pedersen ML, Ironside M, Amemori KI, McGrath CL, Kang MS, Graybiel AM, Pizzagalli DA, Frank MJ. Computational phenotyping of brain-behavior dynamics underlying approach-avoidance conflict in major depressive disorder. PLoS Comput Biol. 2021 May 10;17(5):e1008955. doi: 10.1371/journal.pcbi.1008955. eCollection 2021 May. PMID 33970903
- [Background] Cisler JM, Esbensen K, Sellnow K, Ross M, Weaver S, Sartin-Tarm A, Herringa RJ, Kilts CD. Differential Roles of the Salience Network During Prediction Error Encoding and Facial Emotion Processing Among Female Adolescent Assault Victims. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Apr;4(4):371-380. doi: 10.1016/j.bpsc.2018.08.014. Epub 2018 Sep 11. PMID 30343131
- [Background] Ross MC, Lenow JK, Kilts CD, Cisler JM. Altered neural encoding of prediction errors in assault-related posttraumatic stress disorder. J Psychiatr Res. 2018 Aug;103:83-90. doi: 10.1016/j.jpsychires.2018.05.008. Epub 2018 May 12. PMID 29783079
- [Background] Cisler JM, Tamman AJF, Fonzo GA. Diminished prospective mental representations of reward mediate reward learning strategies among youth with internalizing symptoms. Psychol Med. 2023 Oct;53(14):6910-6920. doi: 10.1017/S0033291723000478. Epub 2023 Mar 7. PMID 36878892
- [Background] Keren H, O'Callaghan G, Vidal-Ribas P, Buzzell GA, Brotman MA, Leibenluft E, Pan PM, Meffert L, Kaiser A, Wolke S, Pine DS, Stringaris A. Reward Processing in Depression: A Conceptual and Meta-Analytic Review Across fMRI and EEG Studies. Am J Psychiatry. 2018 Nov 1;175(11):1111-1120. doi: 10.1176/appi.ajp.2018.17101124. Epub 2018 Jun 20. PMID 29921146
- [Background] Webb CA, Murray L, Tierney AO, Forbes EE, Pizzagalli DA. Reward-related predictors of symptom change in behavioral activation therapy for anhedonic adolescents: a multimodal approach. Neuropsychopharmacology. 2023 Mar;48(4):623-632. doi: 10.1038/s41386-022-01481-4. Epub 2022 Oct 28. PMID 36307561
- [Background] Huys QJ, Pizzagalli DA, Bogdan R, Dayan P. Mapping anhedonia onto reinforcement learning: a behavioural meta-analysis. Biol Mood Anxiety Disord. 2013 Jun 19;3(1):12. doi: 10.1186/2045-5380-3-12. PMID 23782813
- [Background] Hedtke KA, Ruggiero KJ, Fitzgerald MM, Zinzow HM, Saunders BE, Resnick HS, Kilpatrick DG. A longitudinal investigation of interpersonal violence in relation to mental health and substance use. J Consult Clin Psychol. 2008 Aug;76(4):633-47. doi: 10.1037/0022-006X.76.4.633. PMID 18665691
- [Background] Lippard ETC, Nemeroff CB. The Devastating Clinical Consequences of Child Abuse and Neglect: Increased Disease Vulnerability and Poor Treatment Response in Mood Disorders. Am J Psychiatry. 2023 Aug 1;180(8):548-564. doi: 10.1176/appi.ajp.19010020. PMID 37525603
- [Background] Nemeroff CB. Paradise Lost: The Neurobiological and Clinical Consequences of Child Abuse and Neglect. Neuron. 2016 Mar 2;89(5):892-909. doi: 10.1016/j.neuron.2016.01.019. PMID 26938439

DOCUMENTS (2):
  • Study Protocol (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07369115/Prot_000.pdf
  • Informed Consent Form (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07369115/ICF_001.pdf